CLINICAL TRIAL: NCT03652545
Title: Phase I REsearch on Multi-antigen T Cell Infusion Against Neuro-oncologic Disease
Brief Title: Multi-antigen T Cell Infusion Against Neuro-oncologic Disease
Acronym: REMIND
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Catherine Bollard (Other)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Sponsor-Investigator, Catherine Bollard, Director, center for Cancer and Immunology Research, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00010463
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TAA-T (Experimental): Three different dosing schedules will be evaluated.
  Dose Level One: 2 x 107 cells/m2 Dose Level Two: 4 x 107 cells/m2 Dose Level Three: 8 x 107 cells/m2
  Group A patients (DIPG): The first TAA-T dose will be infused any time more than or equal to 14 days after completion of radiotherapy.
  Group B patients (other recurrent/progressive/refractory CNS tumors): TAA-T will be infused any time more than or equal to 14 days after completing most recent course of conventional (non-investigational) therapy for their disease AND after appropriate washout periods as detailed in eligibility criteria.
  Ideally, patients should not receive other systemic antineoplastic agents for at least 42 days after the infusion of TAA-T, although such treatment may be added if deemed critical for patient care by the attending physician.
  Interventions: Biological: TAA-T

INTERVENTIONS:
Biological: TAA-T — Patients with newly diagnosed diffuse intrinsic pontine gliomas DIPGs (Group A) or recurrent, progressive, or refractory non-brainstem CNS malignancies (Group B). The goal of this cell infusion will be to initiate an immune response against brain tumors that includes multiple antigens and may prevent tumor evasion (through decreased expression of a single antigen)

SUMMARY:
This Phase I dose-escalation trial is designed to determine the safety and feasibility of rapidly generated tumor multi-antigen associated specific cytotoxic T lymphocytes (TAA-T) in patients with newly diagnosed diffuse intrinsic pontine gliomas DIPGs (Group A) or recurrent, progressive, or refractory non-brainstem CNS malignancies (Group B).

Pediatric and adult patients who have high-risk CNS tumors known to typically have positivity for one or more Tumor Antigen Associated (TAA) (WT1, PRAME and/or Survivin) will be eligible. TAA-T will all be generated from patient peripheral blood mononuclear cells (PBMC).

Group A patients (DIPG): The first TAA-T dose will be infused any time 14 days or more after completion of radiotherapy.

Group B patients (other recurrent/progressive/refractory CNS tumors): The first TAA-T dose will be infused any time 14 days or more after completing most recent course of conventional (non-investigational) therapy for their disease AND after appropriate washout periods as detailed in eligibility criteria.

DETAILED DESCRIPTION:
This protocol is designed as a phase I dose-escalation study. Three different TAA-T dose levels will be evaluated in each treatment group (A and B) (see below) with 2 to 4 patients enrolled at each dose level.

Dose Level 1: 2 x 107 cells/m2 Dose Level 2: 4 x 107 cells/m2 Dose Level 3: 8 x 107 cells/m2

Two patients will be initially enrolled to the lowest dose level cohort (separately on each arm) and followed for 42 days after initial TAA-T for DLT evaluations. The decision on whether it is safe to escalate to next dose level or not will be made after at least two patients in each dose level have finished their 42-days toxicity follow up after initial TAA-T. If the first two patients have not finished their 42 days follow-up, up to 2 additional incoming patients can be enrolled at the current dose level.

Ideally, patients should not receive other systemic antineoplastic agents for at least 42 days after infusion of TAA-T (for purposes of evaluation), although such treatment may be added if deemed critical for patient care by the attending physician.

Each patient will receive at least one TAA-T infusion and may receive a maximum of 8 subsequent infusions. The first and second infusions will be administered at least 42 days apart then additional infusions will be spaced at least 28 days apart from each other. The expected volume of each infusion is 1 to 10 ml.

If patients with disease have a response of stable disease or better by RANO criteria at the day 28 evaluation after the second infusion OR if they have clinical stability and a clinical assessment of possible pseudoprogression on MRI, they are eligible to receive up to 6 additional infusions of TAA-T at 28 day intervals if available. Each subsequent infusion will be the same as the enrollment dose level (i.e. no subsequent dose escalation). The first and second infusions will be administered at least 42 days apart then additional infusions will be spaced at least 28 days apart from each other. Following the first infusion, if a patient's TAA-T supply is insufficient for subsequent infusions at the enrollment dose level, further treatments may be administered at a lower dose level at the treating physician's discretion.

If patients who are clinically stable are deemed to have likely pseudoprogression at the disease evaluation after the second infusion or on subsequent imaging, then these patients may still be eligible for infusion if serial imaging and clinical assessments demonstrate stability most consistent with pseudoprogression. In these patients, disease assessment after the imaging that first raises the concern for pseudoprogression (potential progressive disease versus pseudoprogression) must be at least stable when compared with the first scan demonstrating pseudoprogression.

ELIGIBILITY:
Inclusion Criteria:

Recipient Procurement Inclusion Criteria

* Diagnosis of high-risk CNS tumors: DIPG, high-grade glioma, medulloblastoma, ependymoma, embryonal tumors, choroid plexus carcinoma, other aggressive CNS malignancies.

  o Group A (newly diagnosed DIPG): Radiographic diagnosis with DIPG defined as tumors with a pontine epicenter and diffuse intrinsic involvement of the pons. For Group A, procurement within the first 12 weeks after completion of radiotherapy is required.
  * Group B: Recurrent, progressive, or refractory disease after standard treatment. Refractory disease includes high-risk tumors with residual disease after completion of standard treatment or tumors with known poor cure rates with standard treatment.
* 6 months to 80 years of age at enrollment
* Karnofsky/Lansky score of ≥ 60%
* Organ function:

  o ANC greater than or equal to750/µL

  o Platelets greater than or equal to 75K

  o Bilirubin less than or equal to 1.5x ULN

  o AST/ALT less than or equal to 5x ULN

  o Serum creatinine less than or equal to 1.0mg/dL or 1.5x ULN for age (whichever is higher)
  * Pulse oximetry > 90% on room air
* Agree to use contraceptive measures during study protocol participation (when age appropriate)
* Patient or parent/guardian capable of providing informed consent
* Available pre-trial tumor tissue (Optional for Group B patients, but highly encouraged. Also optional for Group A)
* Patient deemed to be of sufficient size in order to provide the necessary blood volume for TAA-T generation

Recipient Procurement Exclusion Criteria

* Patients with uncontrolled infections
* Patients with known HIV infection
* Pregnancy** or lactating females
* Prior immunotherapy with an investigational agent within the last 28 days prior to procurement
* Patients with previous history of allogeneic stem cell transplantation (however, patients who have received autologous stem-cell infusions will remain eligible).
* Bulky tumor o Group B - patients who have bulky tumor on imaging are ineligible. These include the following: Tumor with any evidence of uncal herniation or significant midline shift Tumor with a significant brainstem component Patients who are deemed to have overly bulky tumor by the PI of the study

  * Pregnancy assessment on all patients >7 years will be performed. If patient has child bearing potential (per PI/Sub-I discretion), then pregnancy testing will be performed.

Recipient Inclusion Criteria for Initial TAA-T Administration and for Subsequent Infusions

* Steroids < 0.5 mg/kg/day dexamethasone or equivalent
* Karnofsky/Lansky score of greater than or equal to 60%
* Organ function:

  o ANC greater than or equal to750/µL

  o Platelets greater than or equal to 75K
  * Bilirubin less than or equal to 1.5x ULN
  * AST/ALT less than or equal to 5x ULN
  * Serum creatinine less than or equal 1.0mg/dL or 1.5x ULN for age (whichever is higher)
  * Pulse oximetry > 90% on room air
* Patients must have received their last dose of known:

  o Myelosuppressive chemotherapy (including completing radiotherapy for group A patients): greater than or equal to14 days prior to TAA-T infusion or demonstrated count recovery

  o Investigational agent: 28 days prior to TAA-T infusion. For investigational agents that have known adverse events occurring beyond 28 days after administration, this period must be extended beyond the time when new adverse events are known to commonly occur.
  * Biologic agents: 7 days prior to TAA-T infusion. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time when new adverse events are known to commonly occur.
  * Bevacizumab: bevacizumab may be used if clinically indicated in order to control potential pseudoprogression* or inflammation thought to be due to the cellular product. There will not be a standard required washout period for bevacizumab if used for this indication.
  * Surgery: patients must have recovered from all acute effects of prior surgical intervention
* Neurologic status: Patients with neurologic deficits must have deficits that are stable for a minimum of 7 days prior to TAA-T infusion

  * Pseudoprogression is a retrospective assessment that some (or all) noted tumor enlargement by radiographic criteria may reflect immune cell infiltration rather than true tumor progression. This diagnosis is commonly accepted to be retrospectively true if, in the context of clinical stability, radiographic progression plateaus when it would have been expected to progress.

Recipient Exclusion Criteria for Initial and Subsequent TAA-T Infusions

* Patients with uncontrolled infections
* Bulky tumor*** o Group B - patients who have bulky tumor on imaging are not eligible. These include the following: Tumor with evidence of uncal herniation or significant midline shift Tumor with a significant brainstem component Patients who are deemed to have overly bulky tumor by the PI of the study
* Patients who received ATG, Campath or other immunosuppressive T cell monoclonal antibodies within 28 days of TAA-T cell infusion.

Pregnancy** or lactating females

** Pregnancy assessment on all patients >7 years will be performed. If patient has child bearing potential (per PI/Sub-I discretion), then pregnancy testing will be performed.

*** For subsequent infusions, the most recent disease assessments (as obtained per standard of care) will be used to determine eligibility.

Ages: 6 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Product- Adverse Events | Within 42 days of the first TAA-T dose
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.03, change from Baseline Infusion related toxicity at 42 days.

SECONDARY OUTCOMES:
TAA-T responses | 1 year
  Determine the number of patients who respond to tumor associated antigen lymphocytes from base line to one year.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Hwang, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Brain Tumor Institute, Children's National Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No